CLINICAL TRIAL: NCT06612255
Title: A Phase 1, Single Part, Partially Randomised, Open-Label Study to Evaluate the Relative Bioavailability of a Taste-Masked Delafloxacin Powder for Oral Suspension With Oral Delafloxacin Tablet Reference in Healthy Subjects
Brief Title: A Study Comparing the Bioavailability of a Taste-masked Delafloxacin Powder for Oral Suspension With the Delafloxacin Tablet in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study goals not met
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ML-DEL-101-3727-1; 1009679 (Other: Integrated Research Application System (IRAS)); QSC300553 (Other: Quotient Sciences Study Number)
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Delafloxacin; Baxdela; BARDA; Bioavailability; Taste-masked
MeSH Terms: interventions — delafloxacin; WQ 3034

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen A then B: Delafloxacin Tablet then Powder (Experimental): Participants will receive delafloxacin tablet in the fasted state (Regimen A), followed by delafloxacin powder in the fasted state (Regimen B).
  Interventions: Drug: Delafloxacin; Drug: Delafloxacin Powder
- Regimen B then A: Delafloxacin Powder then Tablet (Experimental): Participants will receive delafloxacin powder in the fasted state (Regimen B), followed by delafloxacin tablet in the fasted state (Regimen A).
  Interventions: Drug: Delafloxacin; Drug: Delafloxacin Powder
- Regimen C: Delafloxacin Powder (Experimental): Participants will receive delafloxacin powder in fasted or fed states.
  Interventions: Drug: Delafloxacin Powder
- Regimen D (Optional): Delafloxacin Powder (Experimental): Participants will receive delafloxacin powder in fasted or fed states.
  Interventions: Drug: Delafloxacin Powder

INTERVENTIONS:
Drug: Delafloxacin — Delafloxacin tablet
  Other Names: Baxdela; Quofeni; Delabaxi; RX-3341; ABT-492; ABT-319492; WQ-3034
  Arms: Regimen A then B: Delafloxacin Tablet then Powder; Regimen B then A: Delafloxacin Powder then Tablet
Drug: Delafloxacin Powder — Delafloxacin powder for oral suspension formulation

SUMMARY:
This study will compare the bioavailability of a novel powder for oral suspension formulation of delafloxacin, intended for treatment of community acquired bacterial pneumonia, to that of the licensed delafloxacin oral tablet in healthy adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Must agree to adhere to the protocol-specified contraception requirements.
* Body mass index of 18.0 to 32.0 kilograms (kg)/meter squared as measured at screening.
* Weight ≥50 kg at screening.

Key Exclusion Criteria:

* Any history of hypersensitivity to delafloxacin or any other fluoroquinolones or previous history of tendon disorders related to fluoroquinolone administration.
* History of clinically significant cardiovascular, renal, hepatic, respiratory, or particularly gastrointestinal disease.
* Participant has a medical condition that may adversely affect taste or smell activity including but not limited to mouth ulcers, significant gum disease, and respiratory and/or sinus infection or cold.
* Clinically significant abnormal clinical chemistry, hematology or urinalysis as judged by the Investigator. Participants with Gilbert's Syndrome are not allowed.
* Participants who do not agree to eat a high-fat breakfast.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, Inc.
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the interim decision meeting following dosing of Regimen A and Regimen B, it was decided not to proceed with Regimen C and Regimen D of the study, and subsequently the decision was made to terminate the study early. Therefore, data were only collected for Regimen A and Regimen B.
Groups:
- Regimen A Then B: Delafloxacin Tablet Then Powder: Participants received delafloxacin tablet in a fasted state (Regimen A), followed by delafloxacin powder in a fasted state (Regimen B).
- Regimen B Then A: Delafloxacin Powder Then Tablet: Participants received delafloxacin powder in a fasted state (Regimen B), followed by delafloxacin tablet in a fasted state (Regimen A).
Period: First Intervention
Arm/Group | Regimen A Then B: Delafloxacin Tablet Then Powder | Regimen B Then A: Delafloxacin Powder Then Tablet
Started | 8 | 8
Receive at Least 1 Dose of Study Drug | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (4 Days)
Arm/Group | Regimen A Then B: Delafloxacin Tablet Then Powder | Regimen B Then A: Delafloxacin Powder Then Tablet
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Regimen A Then B: Delafloxacin Tablet Then Powder | Regimen B Then A: Delafloxacin Powder Then Tablet
Started | 8 | 8
Receive at Least 1 Dose of Study Drug | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A Then B: Delafloxacin Tablet Then Powder | Regimen B Then A: Delafloxacin Powder Then Tablet | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (10.3) | 36.0 (14.4) | 35.6 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Mean Concentration Time Curve From Time 0 to 24 Hours Post-dose (AUC0-24) of Delafloxacin Powder Compared to Oral Delafloxacin Tablet
Description: Blood samples were obtained at protocol-specified timepoints. Results reported as nanograms*hour/milliliter (ng*h/mL).
Time Frame: Pre-dose on Day 1, up to 24 hours post-dose
Population: Pharmacokinetic Analysis Set: all participants who received at least 1 dose of study drug and who were evaluable for this outcome measure at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Regimen A: Delafloxacin Tablet: Participants received delafloxacin tablet in a fasted state.
- Regimen B: Delafloxacin Powder: Participants received delafloxacin powder in a fasted state.
Arm/Group | Regimen A: Delafloxacin Tablet | Regimen B: Delafloxacin Powder
Number analyzed (Participants) | 16 | 16
ng*h/mL | 15700 (26.9) | 8120 (33.9)
Statistical Analysis 1: Comparison: Regimen A: Delafloxacin Tablet vs Regimen B: Delafloxacin Powder; Results obtained from mixed effects model of natural log transformed pharmacokinetic parameters including terms for regimen, period and sequence fitted as fixed effects and subject nested within sequence fitted as a random effect; Test type: Other — Ratio (%) of adjusted geometric means with comparison presented as test (powder)/reference (tablet); Fixed Effect Analysis = 51.68, 90% CI 2-sided [45.71 to 58.43]

2. Secondary Outcome: Maximum Observed Concentration (Cmax) of Delafloxacin Powder
Description: Blood samples were obtained at protocol-specified timepoints. Results reported as nanograms/milliliter (ng/mL).
Time Frame: Pre-dose on Day 1, up to 48 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Regimen B: Delafloxacin Powder
Number analyzed (Participants) | 16
ng/mL | 1850 (33.4)

3. Secondary Outcome: Area Under the Curve From Time 0 to the Time of Last Measurable Concentration (AUC0-last) of Delafloxacin Powder
Description: Blood samples were obtained at protocol-specified timepoints. Results reported as ng*h/mL.
Time Frame: Pre-dose on Day 1, up to 48 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Regimen B: Delafloxacin Powder
Number analyzed (Participants) | 16
ng*h/mL | 8450 (33.5)

4. Secondary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant that occurred either before dosing or once an investigational medicinal product (IMP) had been administered, including occurrences which were not necessarily caused by or related to that product. Treatment-emergent adverse events were AEs that commenced during/after the first administration of IMP or commenced before first administration of IMP, that is, a pre-dose AE or existing medical condition, but worsened in intensity during exposure to IMP. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 through Day 6
Population: Safety Analysis Set: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A: Delafloxacin Tablet | Regimen B: Delafloxacin Powder
Number analyzed (Participants) | 16 | 16
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Day 1 through Day 6
Description: All reported safety data based upon the Safety Analysis Set: all participants who received any amount of study drug. During the interim decision meeting following dosing of Regimen A and Regimen B, it was decided not to proceed with Regimen C and Regimen D of the study, and subsequently the decision was made to terminate the study early. Therefore, safety data were only collected for Regimen A and Regimen B.
Arm/Group | Regimen A: Delafloxacin Tablet | Regimen B: Delafloxacin Powder
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Delafloxacin Tablet (N=16) | Regimen B: Delafloxacin Powder (N=16)
Headache (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Catheter site pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Following interim review of the pharmacokinetics and safety data, the decision was made to terminate the study early owing to lower-than-expected exposure levels for delafloxacin powder for oral suspension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT06612255/Prot_001.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT06612255/SAP_002.pdf
  • Informed Consent Form (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT06612255/ICF_000.pdf